CLINICAL TRIAL: NCT00336635
Title: Randomized, Double Blind, Placebo Control Study to Evaluate the Safety and Immunogenicity of CJ-50300 in Healthy Volunteers : Phase I
Brief Title: Safety and Immunogenicity of CJ-50300
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: HK inno.N Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CJ_SPX_101
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Smallpox
Keywords: smallpox, vaccine, immunity
MeSH Terms: conditions — Smallpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cell-culture derived smallpox vaccine

SUMMARY:
The currently available stock of smallpox vaccine would be insufficient in the face of an incident of smallpox attack. Thus, new manufacturing methods for smallpox vaccine is urgently needed because previous manufacturing methods using calf lymph are no longer acceptable in the view of current standards. Recently, CJ corporation in Republic of Korea has developed cell-culture derived smallpox vaccine (CJ-50300) which was manufactured by infecting MRC-5 cells. The aim of this phase 1 clinical trial were to assess safety, reactogenicity, and immunogenicity of CJ-50300.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Korean male and female subjects between 20 and 28 years of age at the time of screening visit.
2. Willing to participate and have signed the informed consent form
3. In good general health, without clinically skin diseases history, physical examination or laboratory test results
4. Hematocrit >33% for women; >38% for men
5. White cell count 3,300-12,000/mm3
6. Total lymphocyte count > 800 cells/mm3

Exclusion Criteria:

1. Diseases or conditions that cause immunodeficiency (For examples; HIV AIDS, leukemia, lymphoma, generalized malignancy, agammaglobulinemia, history of transplantation, therapy with alkylating agents, antimetabolites, radiation, or oral or parenteral corticosteroids).
2. In close physical contact (household or at work) with an individual who has the diseases or conditions that cause immunodeficiency
3. history or present of eczema or atopic dermatitis
4. Allergy or sensitivity to any known components of vaccine or other medicines
5. In close physical contact (household or at work) with an individual who has acute or chronic skin conditions such as dermatitis, exfoliative dermatitis
6. Subjects with inflammatory ophthalmic disease requiring steroid therapy
7. Subjects who are planning for blood donations
8. Autoimmune disease such as lupus erythematosus
9. Subjects who work in medical institution
10. Household contacts with women who are pregnant or breast-feeding
11. Female Subjects who are pregnant or breast-feeding and have positive result by serum pregnancy test or urine pregnancy test, or do not using approved contraceptives such as sterilization, contraceptive ring injectable, combined oral contraceptive pills and barrier contraceptive, combined hormone-based therapy, contraceptive cream, contraceptive jelly, diaphragm or condoms
12. Subjects household member <1 year old or work with children <1 year old
13. Subjects with a known history of Cardiac disease or have three or more of the following risk factors: hyperpiesia, obesity, hyperlipidemia, glucosuria, sclerosis, cerebral arteriosclerosis
14. Receipt of immunoglobulin and steroid within 14 days of vaccination
15. Receipt of investigational research agents within 120 days of vaccination
16. HBsAg seropositive
17. HCV antibody seropositive
18. HIV seropositive
19. Subjects having fever (oral temperature > 38℃) or severe nutrition disorder
20. Blood donation within 12 weeks in advance screening visit
21. Subject who are not suitable to participate in study according to invesigator's judgement

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
safety and immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-don Oh, MD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim SH, Choi SJ, Park WB, Kim HB, Kim NJ, Oh MD, Choe KW. Detailed kinetics of immune responses to a new cell culture-derived smallpox vaccine in vaccinia-naive adults. Vaccine. 2007 Aug 14;25(33):6287-91. doi: 10.1016/j.vaccine.2007.05.044. Epub 2007 Jun 11. PMID 17597266